CLINICAL TRIAL: NCT03675620
Title: Effects of Blood Flow Restriction Training Compared With Standard Rehabilitation in Patients Following Glenoid Labral Repair
Brief Title: Blood Flow Restriction Training Following Glenoid Labral Repair
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left research facility.
Sponsor: Andrews Research & Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1309802
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Glenoid Labrum Tear

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized control trial. After consenting, subjects will be randomized to one of two groups by using a computer generated random number generator.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Investigators recording data and the patients physician will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Rehabilitation (Control Group) (Active Comparator): All participants will perform traditional post-operative shoulder rehabilitation exercises. Participants randomized to this group will begin with lower extremity strengthening exercises (prior to shoulder strengthening) 2-3 times per week for for the first 6 weeks of post-operative care. Standard rehabilitation will continue until discharge.
  Interventions: Other: Standard Rehabilitation
- Blood Flow Restriction (BFR) (Experimental): All participants will perform traditional post-operative shoulder rehabilitation exercises. Participants randomized to the BFR group will begin combining BFR with lower extremity strengthening exercises (prior to shoulder strengthening) 2-3 times per week for the first 6 weeks post-operative care. Standard rehabilitation will continue until discharge.
  Interventions: Device: BFR

INTERVENTIONS:
Device: BFR — Delfi's Personalized Tourniquet System for Blood Flow Restriction will be used with leg extension and leg press exercises. Bilateral thigh cuffs will be applied to the participants and occlusion pressure will be set at 80% of total occlusive pressure as determined by the Doppler sensor. Each participant will perform 4 sets of each exercise (1 set of 30 repetitions followed by 3 sets of 15 repetitions) with resistance of 30% 1-repetition maximum. The pressure will remain through completion of the final set, but not to exceed 5 minutes. One minute rest without tourniquet application will be performed between exercises. Sets and repetitions will remain constant for each participant; however, resistance will be incrementally increased.
  Arms: Blood Flow Restriction (BFR)
Other: Standard Rehabilitation — The control group will perform perform 4 sets of leg extensions and leg press (1 set of 30 repetitions followed by 3 sets of 15 repetitions) with resistance of 30% 1-repetition maximum. Sets and repetitions will remain constant for each participant; however, resistance will be incrementally increased.
  Arms: Standard Rehabilitation (Control Group)

SUMMARY:
The objective of this study is to evaluate the effects of BFR training on patient reported outcome measures and shoulder muscle girth in patients following glenoid labral repair. The investigators hypothesize that participants receiving BFR with rehabilitation will have greater improvements in patient reported outcome measures and shoulder muscle girth than participants who are treated without BFR.

DETAILED DESCRIPTION:
Patients between the ages of 18 and 55 who had a superior labrum anterior to posterior (SLAP) repair, anterior labral repair, anterior capsulorrhaphy, or posterior labral repair will be screened for participation in this study. Participants will be randomized in a 1:1 ratio to receive standard physical therapy with blood flow restriction training or without blood flow restriction. Participants will receive standard of care rehabilitation for labral repair regardless of group assignment. The length of each physical therapy session will be approximately one hour. The BFR and control group will perform leg press and leg extension exercises prior to shoulder strengthening. The resistance for both groups will be set as 30% of one repetition maximum (1-RM). The goal will be for the participants to perform 4 sets of repetitions sequenced 30, 15, 15, 15 of each exercise, if this is not obtainable then the number of set/repetitions will be decreased. The lower extremity strengthening exercises for this study will be performed by all participants beginning at the first physical therapy visit post-surgery. These exercises will be performed at each physical therapy session for 6 consecutive weeks (approximately 2-3 sessions/week). Standard rehabilitation will continue at the conclusion of the 6-week intervention for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Superior labrum anterior to posterior (SLAP) repair, anterior labral repair, anterior capsulorrhaphy, or posterior labral repair
* Willing to complete their post-operative rehabilitation at Andrews Institute Physical Therapy

Exclusion Criteria:

* Patients with prior procedures or significant injuries to the same shoulder will be excluded
* Patients with arthroscopic debridement of labral tears alone
* Patients with concomitant rotator cuff repair surgery
* Patients with Workers' Compensation or automobile insurance claim will be excluded.
* Patients who have a medical history involving any of the following medical conditions will be excluded - uncontrolled hypertension, diabetes, autoimmune disorders, rheumatoid or psoriatic arthritis, multiple sclerosis, peripheral vascular disease, peripheral neuropathy, deep vein thrombosis, pulmonary embolism, myocardial infarction, stroke, blood disorders, disorders requiring immunosuppression, cancer, an ongoing infectious disease, use of steroids, or significant cardiovascular, renal, hepatic or pulmonary disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Change in Pennsylvania Shoulder Score (PENN) | Baseline (prior to surgery), 1 week, 6 weeks, 16 weeks, 20 weeks, discharge from physical therapy, 1-year, and 2-years post-surgery
  The Penn Shoulder Score contains a visual analog scale pain score for pain at rest, pain with everyday activities, and pain with strenuous activities. The maximum possible score is 100 points.

SECONDARY OUTCOMES:
Change in Global Rating of Change (GROC) | Baseline (prior to surgery), 1 week, 6 weeks, 16 weeks, 20 weeks, discharge from physical therapy, 1-year, and 2-years post-surgery
  Survey that assesses participants change in pain overall, since their injury, since their last physical therapy visit, and since the start of physical therapy
Change in Pain Scale | Baseline (prior to surgery), 1 week, 6 weeks, 16 weeks, 20 weeks, discharge from physical therapy, 1-year, and 2-years post-surgery
  Survey assessing current level of pain
Change in Patient Acceptable Symptom State (PASS) | Baseline (prior to surgery), 1 week, 6 weeks, 16 weeks, 20 weeks, discharge from physical therapy, 1-year, and 2-years post-surgery
  Survey utilizing a 2-item question asking participants their opinion of their current state
Change in Single Assessment Numeric Evaluation (SANE) | Baseline (prior to surgery), 1 week, 6 weeks, 16 weeks, 20 weeks, discharge from physical therapy, 1-year, and 2-years post-surgery
  Survey using a visual analog scale to rate current pain
Change in Patient Centered Outcome Questionnaire | Baseline (prior to surgery), 1 week, 6 weeks, 16 weeks, 20 weeks, discharge from physical therapy, 1-year, and 2-years post-surgery
  Survey that assesses pain, fatigue, distress, and interference with daily activities
Change in Shoulder Girth | Baseline (prior to surgery), 1 week, 6 weeks, 16 weeks, 20 weeks, discharge from physical therapy, 1-year, and 2-years post-surgery
  Circumference of the upper arm will be measured with a tape measure

CONTACTS AND LOCATIONS:
Overall Officials: Adam Anz, MD, Principal Investigator — Andrews Institute for Sports Medicine and Orthopaedics
Locations (1):
- Andrews Institute for Orthopaedics & Sports Medicine, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No